CLINICAL TRIAL: NCT02516176
Title: The Feasibility and Efficacy of Induced Lateral Step Treadmill Training to Improve Paretic Limb Stepping Post-Stroke
Brief Title: Sideways Treadmill Training to Improve Paretic Leg Stepping in Persons Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lois Deming Hedman, Associate Professor of Physical Therapy, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU000200161
Record Dates: First submitted 2015-07-22; First posted 2015-08-05 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; cerebral vascular accident; balance; treadmill; falls; hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treadmill Training (Experimental): Paretic leg step training while standing on a treadmill sideways and responding to treadmill being turned on suddenly.
  Interventions: Behavioral: treadmill training

INTERVENTIONS:
Behavioral: treadmill training — Paretic leg step training while standing on a treadmill sideways and responding to treadmill being turned on suddenly.

SUMMARY:
People who are living in the community following a stroke fall frequently. The ability to take a step in response to a balance disturbance helps to prevent falls but stroke survivors tend not to step with their paretic leg in these circumstances. This leaves them vulnerable to falls towards their paretic side. The purpose of this study is to train paretic limb stepping by having individuals stand sideways on a treadmill and respond to sudden accelerations of the treadmill.

DETAILED DESCRIPTION:
Stroke survivors living in the community are at high risk for falling. Falls are considered to be one of the most prevalent post-stroke complications. Fall history in this population has been associated with developing activity limitation, decreased independence and increased fear of falling.

The ability to step in response to an equilibrium disturbance is considered to be critical to prevent a fall. Stroke survivors tend not to step with their paretic limb when their standing equilibrium is perturbed. Training the paretic limb to step in response to perturbations has had limited success in stroke survivors. In response to sagittal plane perturbation training, stroke survivors continued tend to step with their non-paretic leg even when cued or induced to step with paretic leg. This tendency decreases their flexibility to respond to perturbations and also makes it difficult to train the paretic limb.

In contrast, coronal plane perturbations may be a useful way to induce paretic limb stepping. Acceleration and deceleration of a treadmill has been used to train reactive stepping in all directions persons with Parkinson's Disease. Coronal plane perturbations may elicit greater responses from the paretic limb but this has never been investigated in the stroke population.

In this study participants will engage in 6 training sessions over 2-3 weeks. They will stand sideways on the treadmill with their paretic leg towards the front of the treadmill belt, which will be suddenly accelerated for 3 seconds to a predetermined velocity. Participants will perform 80 trials each session under one or more of the following four training conditions.

NON-ENCOURAGED TREADMILL ONLY: These trials are defined as trials when the subject is instructed to respond as necessary to remain on the front half of the treadmill while maintaining their balance without using external supports, but are not given any specific instructions about which limb to use to initiate stepping when the treadmill begins to move.

NON-ENCOURAGED USE TREADMILL PLUS SECONDARY TASK: All the same procedures for non-encouraged use treadmill only trials will be used with the following addition. Just after the subject attains equal weight bearing, the subject will be engaged in a cognitive task to name as many items in a category as they are able. During this time period, the treadmill will be started randomly.

ENCOURAGED USE TREADMILL ONLY TRIALS: These trials are defined as trials where subjects will be instructed to respond as necessary to remain on the front half of the treadmill while maintaining their balance without using external supports AND to initiate stepping with his or her paretic leg when the treadmill begins to move.

ENCOURAGED USE TREADMILL PLUS SECONDARY TASK: All the same procedures for encouraged use treadmill only trials will be used with the following addition. Just after the subject attains equal weight bearing, the subject will be engaged in a cognitive task to name as many items in a category as they are able. During this time period, the treadmill will be started at randomly.

In pilot testing, this protocol has been tolerated by most community dwelling stroke survivors and the encouraged use trials with feedback consistently elicited paretic leg reactive steps.

ELIGIBILITY:
Inclusion Criteria for subjects who have had a stroke:

* at least 18 years old
* a stroke survivor for at least 3 months
* able to understand the testing instructions
* able to walk 10 steps independently without an assistive device
* living in the community (at home in an apartment, condo or house).
* may have a history of one or more strokes but must present with one-sided hemiparesis

Exclusion Criteria for subjects who have had a stroke:

* currently participating in physical therapy for balance and gait-training
* other major musculoskeletal or other neurological disorders
* residing in skilled nursing or assisted living facilities.

Exclusion criteria for subjects who have not had a stroke:

* other major musculoskeletal or neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance in the Four Square Step Test | change from baseline at 3 weeks - immediately following the training sessions
  The FSST is a timed test that assesses a person's ability to step forwards, sideways, and backwards over canes that are placed on the floor

CONTACTS AND LOCATIONS:
Overall Officials: Lois D Hedman, DSc PT, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No